CLINICAL TRIAL: NCT02396940
Title: Three-dimensional High-definition (3DHD) Laparoscopy Versus Two-dimensional High-definition (2DHD) Laparoscopy in Inguinal Hernia Repair.
Brief Title: 3D HD Versus 2D HD in Laparoscopic Inguinal Hernia Repair: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Fergo, Miss, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3D_vs_2D_ing
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Hernia, Inguinal; Hernia
Keywords: 3D; Three-dimensional; Laparoscopy; Inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2D HD laparoscopy (Placebo Comparator): Elective laparoscopic inguinal hernia repair performed with the use of Olympus ENDOEYE FLEX in the 2DHD viewing mode
  Interventions: Device: 2D HD laparoscopy
- 3D HD laparoscopy (Active Comparator): Elective laparoscopic cholecystectomy performed with the use of Olympus ENDOEYE FLEX in the 3DHD viewing mode
  Interventions: Device: 3D HD laparoscopy

INTERVENTIONS:
Device: 3D HD laparoscopy — Olympus 3D laparoscopy ENDOEYE FLEX in high definition with the use of passive, polarizing glasses.
  Other Names: Olympus 3D ENDOEYE FLEX
  Arms: 3D HD laparoscopy
Device: 2D HD laparoscopy — Placebo
  Arms: 2D HD laparoscopy

SUMMARY:
The aim of this study is to compare 3D-laparoscopy versus 2D-laparoscopy with the use of HD resolution in inguinal hernia repair in terms of error rating, performance time and subjective assessment.

DETAILED DESCRIPTION:
Experimental studies have shown that even experienced surgeons gain from stereoscopy when solving both easy and complex tasks. Inguinal hernia repair is a specialist operation and the large flow makes this type of operation suitable for exploring any advantage of three-dimensional laparoscopy for the experienced surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective inguinal hernia repair (out-patient treatment)

Exclusion Criteria:

* Previous lower abdominal surgery
* ASA-score 3 or above

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of errors during the dissection of the hernia sac | Expected duration: 20 minutes
  The unedited videos of the operations will be assessed according to GERT (Generic Error Rating Tool) by three surgeons, blinded to which optical modalities is used during the operations as done in a previous pilot study.

SECONDARY OUTCOMES:
Duration of the dissection of the hernia sac. | Expected duration: 20 minutes
Duration of surgery | Expected duration: 1 hour
The need for conversion to open surgery | intraoperative, expected duration of surgery: 1 hour
Estimated blood loss in ml | intraoperative, expected duration of surgery: 1 hour
Intraoperative complications | intraoperative, expected duration of surgery: 1 hour
Assessment of fatigue and perceived exertion | an expected average of 15 minutes before and after the operation
  Subjective assessment. The surgeon will fill out questionnaires and scales
Evaluation of the optical modality and mental load assessment | an expected average of 15 minutes after the operation
  Subjective assessment. The surgeon will fill out questionnaires and scales

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Fergo, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No